CLINICAL TRIAL: NCT03401944
Title: Effects of Total Parenteral Nutrition on Skeletal Muscle Genomics.
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Göteborg University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: MB1+2
Record Dates: First submitted 2017-12-21; First posted 2018-01-17 (Actual); Last update posted 2018-01-23 (Actual); Status verified 2018-01

CONDITIONS: Wasting;Muscle(S)
MeSH Terms: conditions — Muscular Atrophy | interventions — Parenteral Nutrition

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Total Parenteral Nutrition (TPN) (Active Comparator): Overnight infusion of Parenteral Nutrition supplied in all-in one bag -format. Infusion-rate of 0.16 gram Nitrogen/kg/day.
  Interventions: Drug: TPN
- Control (saline infusion) (Placebo Comparator): Overnight infusion of physiological saline at the same infusion-rate; ml/kg as intervention (TPN).
  Interventions: Other: Control

INTERVENTIONS:
Drug: TPN
  Other Names: TPN infusion
  Arms: Total Parenteral Nutrition (TPN)
Other: Control
  Other Names: Physiological saline infusion
  Arms: Control (saline infusion)

SUMMARY:
The study investigates effects related to muscle protein metabolism at provision of Total Parenteral nutrition.

DETAILED DESCRIPTION:
Randomized study investigating alterations in muscle protein metabolism at provision of parenteral nutrition. The study uses a genomic/transcriptomic/proteomic approach to evaluate factors related to activation of skeletal muscle protein synthesis. Patients scheduled for major gastrointestinal surgery are included. Muscle specimens are collected during surgery.

ELIGIBILITY:
Inclusion Criteria:

* Major gastrointestinal surgery
* Assumed need of post-operative artificial nutrition.

Exclusion Criteria:

* Insulin dependent diabetes
* Steroid medication

Ages: 20 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Actual)
Dates: Start 2005-01-01 (Actual); Primary Completion 2014-12-31 (Actual); Study Completion 2014-12-31 (Actual)

PRIMARY OUTCOMES:
Muscle protein metabolism | Single evaluation point at 12-14 hours following the start of overnight infusion.
  Alterations in muscle protein metabolism will be assessed by various standard techniques for gene and protein expression. Combined measurements of cell-signaling molecules representing anabolic and catabolic signaling pathways will be evaluated in relation to transcription of muscle myosin proteins.

CONTACTS AND LOCATIONS:
Overall Officials: Kent Lundholm, Principal Investigator — Department of Surgery, University of Gothenburg
Locations (1):
- Department of Surgery, Gothenburg, Sweden